CLINICAL TRIAL: NCT04675177
Title: Sclerotherapy With Polidocanol Foam Versus Hemorrhoidal Artery Ligation With Recto Anal Repair in the Treatment of Second and Third-grade Hemorrhoidal Disease: a Prospective Study
Brief Title: Polidocanol Foam VS Artery Ligation in Hemorrhoidal Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Paulo Sérgio Durão Salgueiro, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 514741899
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Sclerotherapy; polidocanol foam; Doppler-guided hemorrhoidal artery ligation
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: Prospective, unicentric study (Centro Hospitalar Universitário do Porto (CHUP)) which is aimed to compare the efficacy and safety of the treatment techniques in patients with hemorrhoidal disease grade II and III.
  Patients referred to consultation were randomly allocated to one of the two treatments (polidocanol foam sclerotherapy and hemorrhoid artery ligation +- rectoanal repair).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polidocanol foam sclerotherapy (Active Comparator): Patients submitted to polidocanol foam sclerotherapy
  Interventions: Drug: Polidocanol foam sclerotherapy
- Doppler-guided hemorrhoidal artery ligation (Active Comparator): Patients submitted to doppler-guided hemorrhoidal artery ligation
  Interventions: Procedure: Doppler-guided hemorrhoidal artery ligation

INTERVENTIONS:
Drug: Polidocanol foam sclerotherapy — i. Patients underwent preparation, two hours before the intervention, with cleaning enema (Disodium phosphate). No antibiotic prophylaxis was prescribed.
  ii. Preparation of the polidocanol (Aethoxysklerol 3%) foam according to Tessari technique immediately before application, so that the "microbubbles" of the foam did not disintegrate; iii. The procedure was performed in the medical office. Application according to the Blanchard technique through a disposable transparent anoscope, in jackknife position, using a 20mL disposable syringe of the mixture (polidocanol + air) and a reusable 10 cm syringe extender adapted to an intravenous needle; iv. Patients were treated in a maximum of 3 sessions, at 3 weeks intervals; v. Maximum dose per treatment session of 20mL of mixture of 4mL of polidocanol 3% with 16mL of air; i. In each session, the sclerosant was injected in one or more hemorroidary cushion;
  Other Names: Aethoxysklerol 3%)
  Arms: Polidocanol foam sclerotherapy
Procedure: Doppler-guided hemorrhoidal artery ligation — i. Patients underwent preparation with cleaning enema (Disodium phosphate). No antibiotic prophylaxis was prescribed.
  ii. The procedure was performed in the operating room of an outpatient surgery unit, under regional anestesia.
  iii. A proctoscope with a Doppler transducer in its tip was introduced inside the anal canal to search for the superior rectal artery.
  iv. Each branch was ligated with suture above the dentate line. The device was rotated slowly in clockwise direction to locate further arteries at that level.
  v. Rectoanal repair consisted in a continuous running suture was applied longitudinally just over every prolapsed hemorrhoid.
  Other Names: HAL-RAR
  Arms: Doppler-guided hemorrhoidal artery ligation

SUMMARY:
Background: Hemorrhoidal disease is extremely frequent in the adult population and, as a benign pathology, the treatment should be guided by the patient's symptoms. Treatment of hemorrhoidal disease includes a conservative approach, office-based treatments and surgery.

This study is aimed to evaluate and compare the efficacy and safety of the treatment of hemorrhoidal disease with non-surgical office-based method polidocanol foam sclerotherapy (SP) and the surgical technique doppler-guided hemorrhoidal artery ligation with recto-anal repair.

Methods: Prospective, unicentric study including patients with symptomatic hemorrhoidal disease grade II and III refractory to conservative therapy, submitted either to SP (n=24) or to HAL-RAR procedure (n=21), during a recruitment period of 6 months.

Patients were evaluated for efficacy (Sodergren's scale of symptoms and severity of bleeding) and safety (complications and implication in personal and professional life), up to one month after treatment. In follow-up period (6 months) participants were evaluated for hemorrhoidal disease recurrence.

DETAILED DESCRIPTION:
INTRODUCTION:

Instrumental office-based procedures are usually indicated for internal hemorrhoidal disease grade I and II which are refractory to conservative medical treatments and in selected cases of grade III hemorrhoidal disease. Despite being invasive, these techniques are more conservative than surgical treatments and are also effective. The primary goals are to decrease the amount of redundant tissue, reduce vascularity, and affix the hemorrhoidal cushions to minimize prolapse. Office-based procedures include rubber band ligation (RBL), sclerotherapy (liquid and foam agents), infrared photocoagulation, cryotherapy, radiofrequency ablation among others.

Hemorrhoidal sclerosis is a procedure indicated to treat grade I and II hemorrhoidal disease. It has also been used in the treatment of internal grade III hemorrhoidal disease, but there are limited data on its efficacy. Performed through an anoscope and according to Blanchard technique, internal hemorrhoids are located and injected with a sclerosant material into the submucosa at the base of the hemorrhoid, above the anterolateral line. The sclerosant subsequently causes an inflammatory response and fibrosis that interrupts the vascular blood supply. A variety of sclerosants have been used including ethanolamine, quinine, hypertonic saline, aluminum potassium sulfate and tannic acid (ALTA), and 5% phenol in oil. Recently, a new sclerosing agent, polidocanol, started to be employed in the treatment of hemorrhoidal disease. It is a nonionic detergent and consists of a hydrophilic polyethylene oxide chain combined with hydrophobic aliphatic dodecyl alcohol. When injected into varicose veins, polidocanol damages the endothelium of blood vessels, allowing platelets to aggregate. Eventually, a dense network of platelets, cellular debris, and fibrin occludes the vessel, which is subsequently replaced with connective fibrous tissue. In addition to the treatment of hemorrhoidal disease, polidocanol is used for sclerotherapy of varicose veins of the lower extremities and for the treatment of esophageal varices. The advantages of this sclerosing agent include a highly satisfactory efficiency, a low necrotic potential, and a good general tolerance. At the same time, it has a local anesthetic effect which permits almost painless sclerotherapy. Nevertheless, its use is contraindicated in patients with acute thromboembolic diseases and in those with allergy to the drug. Polidocanol can be used in its liquid or foam form. It has been proved the foam formulation allows for greater efficacy, since it requires lower doses of sclerosant agent. This is because the sclerotic effect is maximized by increasing the contact surface area with varices walls. This foam is previously prepared according to the Tessari's method, in which two 10 mL syringes are connected by a 3-way stopcock. The syringes contain air and a sclerosing agent (3% polydocanol), with a ratio of 4:1, respectively, and twenty passages from one syringe to the other are made in order to obtain a sclerosing foam. Several studies reported the efficacy of the use of sclerotherapy with liquid polidocanol in hemorrhoidal disease. Specifically for the treatment of grade I hemorrhoids, there is one study showing the superiority of polidocanol foam compared to its liquid formulation. However, there's a lack of research about its use in hemorrhoidal disease other than grade I. The most common complications of sclerotherapy include minor discomfort or bleeding. Although it is a very safe treatment option, some serious side effects, including erectile dysfunction and urinary retention, have been reported. The proper injection technique of sclerosant is essential to avoid complications such as mucosal ulceration or necrosis, prostatic abscess and retroperitoneal sepsis. Sclerotherapy is a valid alternative when conservative therapy has failed. Moreover, this procedure can also be used for the treatment of patients whose hemorrhage is the main symptom, for patients on antithrombotic medication, as well as cirrhotic and immunocompromised patients.

Surgical treatment is reserved for refractory cases to nonsurgical approaches, grade IV or mixed hemorrhoidal disease (internal and external components), symptomatic hemorrhoidal disease with concomitant anorectal pathology and lastly if it's the patient's choice. Although surgical approach is apparently more effective than instrumental treatment, it is also associated with substantial postsurgical morbidity, particularly postoperative pain and limitation in day-life activities. Several surgical methods have been described including open and closed hemorrhoidectomy, doppler guided hemorrhoidal artery ligation (HAL) and hemorrhoidectomy stapler. The choice of each method should consider the grade of hemorrhoidal disease and the predominant symptoms of the patient, together with the experience of the center.

HAL technique involves the use of Doppler ultrasound and a specialized anoscope. The principles include the use of a Doppler probe to identify the six main feeding arteries within the anal canal and their ligation with absorbable suture above the dentate line, therefore associated with less pain. Finally, plication of redundant hemorrhoidal mucosa is performed (if there is hemorrhoidal or muco-hemorrhoidal prolapse), known as recto-anal-repair (RAR), mucopexy or hemorrhoidopexy. The aim of this recent surgical procedure is to treat patients' symptoms without tissue destruction. Early results of HAL were promising, with lower pain scores than hemorrhoidectomy, and relief of bleeding and tissue prolapse in over 90% of patients. Since then, several randomized clinical trials have been performed with mixed results. Currently, HAL remains a viable approach to multicolumn internal hemorrhoids. However, the short-term benefits regarding postoperative pain have recently not been as remarkable as in the earlier studies. Also, there has been a progressive increase in long term recurrence rates, especially for grade III and IV hemorrhoids.

Some studies have been conducted with the purpose of comparing the efficacy of nonsurgical office-based treatments with surgical ones.

A multicentric, open-label, randomized controlled trial, compared RBL and HAL, revealing higher efficacy of the surgical procedure. If, however, RBL is considered a course of treatment involving repeat banding, the procedures are equally effective. Besides, HAL was proved to be more painful than RBL. Another study comparing infrared photocoagulation with HAL showed that both procedures are minimally invasive and associated with minimal discomfort, but HAL is more effective than infrared photocoagulation in controlling symptoms of hemorrhoids. There has been no comparative studies between polidocanol foam sclerotherapy and hemorrhoidal artery ligation, to date.

Therefore, the purpose of the present study is to evaluate and compare the safety and efficacy of the treatment of hemorrhoidal disease with polidocanol foam sclerotherapy and HAL-RAR.

METHODS:

Prospective, unicentric study (Centro Hospitalar Universitário do Porto) which is aimed to compare the efficacy and safety of the treatment techniques in patients with hemorrhoidal disease grade II and III.

Patients referred were randomly allocated to one of the two treatments considered in this study (SP and HAL-RAR).

All participants should have had prior endoscopic study, at least sigmoidoscopy, or total colonoscopy if they were older than 50 years or younger, with a family history of colorectal cancer, colon adenomas, or suspected inflammatory bowel disease.

Only patients who agreed to informed consent were included, after a clear explanation of the type of study and the intervention that was going to be made.

In screening visits, demographic and anthropometric data (such as age, sex, weight and height, education and employment status) were collected, as well as grade of hemorrhoidal disease. Baseline questionnaires were used to assess Sodergren's scale of symptoms and the severity of bleeding.

Informed consent and an information brochure, explaining the study and adequate dietary and behavioral care, were provided. Additionally, all participants were given a direct contact for any doubts and notification of complications, in which case additional observation should be made.

When office-based treatment was performed, an intervention period was considered, in which patients were observed at 3-week intervals (the required number of sessions, maximum of 3, depended on the clinical response - if 3 weeks after the previous treatment, the participant scored zero points in the Sodergren scale and had a hemorrhage grade ≤1, he was not a candidate for additional instrumental therapy.).

Surgical treatment was performed only once. One month after this intervention period, Sodergren's scale of symptoms and severity of bleeding were reevaluated. In addition, complications registry, and implication in personal and professional life, measured in number of work-loss days, if applied, were also assessed. Patients was followed-up every 3 months for total of 6 months for evaluation of hemorrhoidal disease symptoms recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with symptomatic hemorrhoidal disease grade II and III (Goligher's classification)
* Refractory to conservative therapy (dietary modification, intestinal transit modifiers, topical and phlebotonic medications) for a period of not less than 4 weeks

Exclusion Criteria:

* Cirrhosis
* Pregnant or breast-feeding women
* Known allergy to polidocanol
* Another perianal disease that can cause symptoms similar to hemorrhoidal disease
* Colorectal malignancy
* Concomitant presence of external hemorrhoidal disease and/or hemorrhoidal thrombosis - - Office or surgical treatment for hemorrhoids within 6 months prior to inclusion
* Antiplatelet or hypocoagulant medication
* Hematological disorders
* Immunosuppressive states
* Inflammatory bowel disease
* Patients unable to have general or spinal anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Therapeutic success | 3 months
  Efficacy indicator composed by Sodergren score and bleeding grade:
  * Complete (Sodergren score = 0 and bleeding grade <= 1);
  * Partial (Sodergren score > 0 and bleeding grade > 1 but, at least, one of them with improvement, regarding the initial score, and none of them worse);
  * Therapeutic failure (participants that, one month after the last instrumental treatment or one month after surgery, worsened or maintained the initial Sodergren score and bleeding grade);
Safety evaluation | 3 Months
  Record of complications resulting from the therapy:
  * Mild (e.g. pain/discomfort, pruritus, bleeding grade 1)
  * Moderate (e.g., external hemorrhoidal thrombosis, bleeding without hemodynamic instability, no blood transfusion, no need for haemostasis or urgent surgery): do not endanger the patient's life or leave long term sequelae;
  * Severe (e.g. sepsis, Fournier's gangrene, perineal abscess, bleeding with hemodynamic instability, transfusional need or urgent surgery, sexual impotence in man): they put the patient's life at risk.

SECONDARY OUTCOMES:
Professional life implications | 3 months
  Implications in professional life were measured in number of work-loss days
Personal life implications | 3 months
  Outcome assessed with some simple yes-no questions (eg: personal and family relationships, sexual activity, physical exercise, social and civic activities), and if at least one of them was answered affirmatively, we considered treatment had significant impact in patient's personal life.
Number of treatment sessions | 3 months
  Number of instrumental treatment sessions required
Recurrence | 6 Months
  Evaluation of symptoms recurrence during de follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Salgueiro, MD, Principal Investigator — Centro Hospitalar Universitário do Porto
Locations (1):
- Centro Hospitalar Universitário do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Study data can shared upon justified request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Justified request (investigation, meta-analysis, medical education)

REFERENCES:
- [Background] Sun Z, Migaly J. Review of Hemorrhoid Disease: Presentation and Management. Clin Colon Rectal Surg. 2016 Mar;29(1):22-9. doi: 10.1055/s-0035-1568144. PMID 26929748
- [Background] Sneider EB, Maykel JA. Diagnosis and management of symptomatic hemorrhoids. Surg Clin North Am. 2010 Feb;90(1):17-32, Table of Contents. doi: 10.1016/j.suc.2009.10.005. PMID 20109630
- [Background] Rakinic J, Poola VP. Hemorrhoids and fistulas: new solutions to old problems. Curr Probl Surg. 2014 Mar;51(3):98-137. doi: 10.1067/j.cpsurg.2013.11.002. Epub 2013 Nov 25. PMID 24606821
- [Background] Lohsiriwat V. Hemorrhoids: from basic pathophysiology to clinical management. World J Gastroenterol. 2012 May 7;18(17):2009-17. doi: 10.3748/wjg.v18.i17.2009. PMID 22563187
- [Background] Lohsiriwat V. Approach to hemorrhoids. Curr Gastroenterol Rep. 2013 Jul;15(7):332. doi: 10.1007/s11894-013-0332-6. PMID 23715885
- [Background] Peery AF, Sandler RS, Galanko JA, Bresalier RS, Figueiredo JC, Ahnen DJ, Barry EL, Baron JA. Risk Factors for Hemorrhoids on Screening Colonoscopy. PLoS One. 2015 Sep 25;10(9):e0139100. doi: 10.1371/journal.pone.0139100. eCollection 2015. PMID 26406337
- [Background] Faccini M, Zuccon W, Caputo P, Gavezzoli D, Manelli A, Bonandrini L. [Hemorrhoids: epidemiology and correlation with chronic constipation]. Ann Ital Chir. 2001 May-Jun;72(3):337-9; discussion 340. Italian. PMID 11765352
- [Background] Pigot F, Siproudhis L, Allaert FA. Risk factors associated with hemorrhoidal symptoms in specialized consultation. Gastroenterol Clin Biol. 2005 Dec;29(12):1270-4. doi: 10.1016/s0399-8320(05)82220-1. PMID 16518286
- [Background] Riss S, Weiser FA, Schwameis K, Riss T, Mittlbock M, Steiner G, Stift A. The prevalence of hemorrhoids in adults. Int J Colorectal Dis. 2012 Feb;27(2):215-20. doi: 10.1007/s00384-011-1316-3. Epub 2011 Sep 20. PMID 21932016
- [Background] Johanson JF, Sonnenberg A. The prevalence of hemorrhoids and chronic constipation. An epidemiologic study. Gastroenterology. 1990 Feb;98(2):380-6. doi: 10.1016/0016-5085(90)90828-o. PMID 2295392
- [Background] Lohsiriwat V. Treatment of hemorrhoids: A coloproctologist's view. World J Gastroenterol. 2015 Aug 21;21(31):9245-52. doi: 10.3748/wjg.v21.i31.9245. PMID 26309351
- [Background] Hollingshead JR, Phillips RK. Haemorrhoids: modern diagnosis and treatment. Postgrad Med J. 2016 Jan;92(1083):4-8. doi: 10.1136/postgradmedj-2015-133328. Epub 2015 Nov 11. PMID 26561592
- [Background] Qureshi WA. Office management of hemorrhoids. Am J Gastroenterol. 2018 Jun;113(6):795-798. doi: 10.1038/s41395-018-0020-0. No abstract available. PMID 29487411
- [Background] Pucher PH, Qurashi M, Howell AM, Faiz O, Ziprin P, Darzi A, Sodergren MH. Development and validation of a symptom-based severity score for haemorrhoidal disease: the Sodergren score. Colorectal Dis. 2015 Jul;17(7):612-8. doi: 10.1111/codi.12903. PMID 25603811
- [Background] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751
- [Background] Park SK, Ko BM, Goong HJ, Seo JY, Lee SH, Baek HL, Lee MS, Park DI. Short health scale: A valid measure of health-related quality of life in Korean-speaking patients with inflammatory bowel disease. World J Gastroenterol. 2017 May 21;23(19):3530-3537. doi: 10.3748/wjg.v23.i19.3530. PMID 28596689
- [Background] Sandler RS, Peery AF. Rethinking What We Know About Hemorrhoids. Clin Gastroenterol Hepatol. 2019 Jan;17(1):8-15. doi: 10.1016/j.cgh.2018.03.020. Epub 2018 Mar 27. PMID 29601902
- [Background] Jacobs D. Clinical practice. Hemorrhoids. N Engl J Med. 2014 Sep 4;371(10):944-51. doi: 10.1056/NEJMcp1204188. No abstract available. PMID 25184866
- [Background] Ganz RA. The evaluation and treatment of hemorrhoids: a guide for the gastroenterologist. Clin Gastroenterol Hepatol. 2013 Jun;11(6):593-603. doi: 10.1016/j.cgh.2012.12.020. Epub 2013 Jan 16. No abstract available. PMID 23333220
- [Background] Iyer VS, Shrier I, Gordon PH. Long-term outcome of rubber band ligation for symptomatic primary and recurrent internal hemorrhoids. Dis Colon Rectum. 2004 Aug;47(8):1364-70. doi: 10.1007/s10350-004-0591-2. PMID 15484351
- [Background] Cocorullo G, Tutino R, Falco N, Licari L, Orlando G, Fontana T, Raspanti C, Salamone G, Scerrino G, Gallo G, Trompetto M, Gulotta G. The non-surgical management for hemorrhoidal disease. A systematic review. G Chir. 2017 Jan-Feb;38(1):5-14. doi: 10.11138/gchir/2017.38.1.005. PMID 28460197
- [Background] Albuquerque A. Rubber band ligation of hemorrhoids: A guide for complications. World J Gastrointest Surg. 2016 Sep 27;8(9):614-620. doi: 10.4240/wjgs.v8.i9.614. PMID 27721924
- [Background] Acheson AG, Scholefield JH. Management of haemorrhoids. BMJ. 2008 Feb 16;336(7640):380-3. doi: 10.1136/bmj.39465.674745.80. No abstract available. PMID 18276714
- [Background] Song SG, Kim SH. Optimal treatment of symptomatic hemorrhoids. J Korean Soc Coloproctol. 2011 Dec;27(6):277-81. doi: 10.3393/jksc.2011.27.6.277. Epub 2011 Dec 31. PMID 22259741
- [Background] Hachiro Y, Kunimoto M, Abe T, Kitada M, Ebisawa Y. Aluminum potassium sulfate and tannic acid (ALTA) injection as the mainstay of treatment for internal hemorrhoids. Surg Today. 2011 Jun;41(6):806-9. doi: 10.1007/s00595-010-4386-x. Epub 2011 May 28. PMID 21626327
- [Background] Hussar DA, Stevenson T. New drugs: Denosumab, dienogest/estradiol valerate, and polidocanol. J Am Pharm Assoc (2003). 2010 Sep-Oct;50(5):658-62. doi: 10.1331/JAPhA.2010.10536. No abstract available. PMID 20833626
- [Background] Moser KH, Mosch C, Walgenbach M, Bussen DG, Kirsch J, Joos AK, Gliem P, Sauerland S. Efficacy and safety of sclerotherapy with polidocanol foam in comparison with fluid sclerosant in the treatment of first-grade haemorrhoidal disease: a randomised, controlled, single-blind, multicentre trial. Int J Colorectal Dis. 2013 Oct;28(10):1439-47. doi: 10.1007/s00384-013-1729-2. Epub 2013 Jun 18. PMID 23775099
- [Background] Yuksel BC, Armagan H, Berkem H, Yildiz Y, Ozel H, Hengirmen S. Conservative management of hemorrhoids: a comparison of venotonic flavonoid micronized purified flavonoid fraction (MPFF) and sclerotherapy. Surg Today. 2008;38(2):123-9. doi: 10.1007/s00595-007-3582-9. Epub 2008 Feb 1. PMID 18239868
- [Background] Nastasa V, Samaras K, Ampatzidis Ch, Karapantsios TD, Trelles MA, Moreno-Moraga J, Smarandache A, Pascu ML. Properties of polidocanol foam in view of its use in sclerotherapy. Int J Pharm. 2015 Jan 30;478(2):588-96. doi: 10.1016/j.ijpharm.2014.11.056. Epub 2014 Nov 26. PMID 25433198
- [Background] Tessari L, Cavezzi A, Frullini A. Preliminary experience with a new sclerosing foam in the treatment of varicose veins. Dermatol Surg. 2001 Jan;27(1):58-60. PMID 11231246
- [Background] Cavezzi A, Tessari L. Foam sclerotherapy techniques: different gases and methods of preparation, catheter versus direct injection. Phlebology. 2009 Dec;24(6):247-51. doi: 10.1258/phleb.2009.009061. PMID 19952380
- [Background] Scaglia M, Delaini GG, Destefano I, Hulten L. Injection treatment of hemorrhoids in patients with acquired immunodeficiency syndrome. Dis Colon Rectum. 2001 Mar;44(3):401-4. doi: 10.1007/BF02234740. PMID 11289287
- [Background] Clinical Practice Committee, American Gastroenterological Association. American Gastroenterological Association medical position statement: Diagnosis and treatment of hemorrhoids. Gastroenterology. 2004 May;126(5):1461-2. doi: 10.1053/j.gastro.2004.03.001. PMID 15131806
- [Background] Conaghan P, Farouk R. Doppler-guided hemorrhoid artery ligation reduces the need for conventional hemorrhoid surgery in patients who fail rubber band ligation treatment. Dis Colon Rectum. 2009 Jan;52(1):127-30. doi: 10.1007/DCR.0b013e3181973639. PMID 19273967
- [Background] Ohning GV, Machicado GA, Jensen DM. Definitive therapy for internal hemorrhoids--new opportunities and options. Rev Gastroenterol Disord. 2009 Winter;9(1):16-26. PMID 19367214
- [Background] Peng BC, Jayne DG, Ho YH. Randomized trial of rubber band ligation vs. stapled hemorrhoidectomy for prolapsed piles. Dis Colon Rectum. 2003 Mar;46(3):291-7; discussion 296-7. doi: 10.1007/s10350-004-6543-z. PMID 12626901
- [Background] Watson AJ, Bruhn H, MacLeod K, McDonald A, McPherson G, Kilonzo M, Norrie J, Loudon MA, McCormack K, Buckley B, Brown S, Curran F, Jayne D, Rajagopal R, Cook JA; eTHoS study group. A pragmatic, multicentre, randomised controlled trial comparing stapled haemorrhoidopexy to traditional excisional surgery for haemorrhoidal disease (eTHoS): study protocol for a randomised controlled trial. Trials. 2014 Nov 11;15:439. doi: 10.1186/1745-6215-15-439. PMID 25388563
- [Background] Yano T, Asano M, Tanaka S, Oda N, Matsuda Y. Prospective study comparing the new sclerotherapy and hemorrhoidectomy in terms of therapeutic outcomes at 4 years after the treatment. Surg Today. 2014 Mar;44(3):449-53. doi: 10.1007/s00595-013-0564-y. Epub 2013 Mar 30. PMID 23543083
- [Background] Yeo D, Tan KY. Hemorrhoidectomy - making sense of the surgical options. World J Gastroenterol. 2014 Dec 7;20(45):16976-83. doi: 10.3748/wjg.v20.i45.16976. PMID 25493010
- [Background] Morinaga K, Hasuda K, Ikeda T. A novel therapy for internal hemorrhoids: ligation of the hemorrhoidal artery with a newly devised instrument (Moricorn) in conjunction with a Doppler flowmeter. Am J Gastroenterol. 1995 Apr;90(4):610-3. PMID 7717320
- [Background] Ratto C. THD Doppler procedure for hemorrhoids: the surgical technique. Tech Coloproctol. 2014 Mar;18(3):291-8. doi: 10.1007/s10151-013-1062-3. Epub 2013 Sep 12. PMID 24026315
- [Background] Hoyuela C, Carvajal F, Juvany M, Troyano D, Trias M, Martrat A, Ardid J, Obiols J. HAL-RAR (Doppler guided haemorrhoid artery ligation with recto-anal repair) is a safe and effective procedure for haemorrhoids. Results of a prospective study after two-years follow-up. Int J Surg. 2016 Apr;28:39-44. doi: 10.1016/j.ijsu.2016.02.030. Epub 2016 Feb 10. PMID 26876958
- [Background] Giordano P, Overton J, Madeddu F, Zaman S, Gravante G. Transanal hemorrhoidal dearterialization: a systematic review. Dis Colon Rectum. 2009 Sep;52(9):1665-71. doi: 10.1007/DCR.0b013e3181af50f4. PMID 19690499
- [Background] De Nardi P, Capretti G, Corsaro A, Staudacher C. A prospective, randomized trial comparing the short- and long-term results of doppler-guided transanal hemorrhoid dearterialization with mucopexy versus excision hemorrhoidectomy for grade III hemorrhoids. Dis Colon Rectum. 2014 Mar;57(3):348-53. doi: 10.1097/DCR.0000000000000085. PMID 24509458
- [Background] Denoya PI, Fakhoury M, Chang K, Fakhoury J, Bergamaschi R. Dearterialization with mucopexy versus haemorrhoidectomy for grade III or IV haemorrhoids: short-term results of a double-blind randomized controlled trial. Colorectal Dis. 2013;15(10):1281-8. doi: 10.1111/codi.12303. PMID 23711288
- [Background] Elmer SE, Nygren JO, Lenander CE. A randomized trial of transanal hemorrhoidal dearterialization with anopexy compared with open hemorrhoidectomy in the treatment of hemorrhoids. Dis Colon Rectum. 2013 Apr;56(4):484-90. doi: 10.1097/DCR.0b013e31827a8567. PMID 23478616
- [Background] Giamundo P. Advantages and limits of hemorrhoidal dearterialization in the treatment of symptomatic hemorrhoids. World J Gastrointest Surg. 2016 Jan 27;8(1):1-4. doi: 10.4240/wjgs.v8.i1.1. PMID 26843909
- [Background] Brown SR, Tiernan JP, Watson AJM, Biggs K, Shephard N, Wailoo AJ, Bradburn M, Alshreef A, Hind D; HubBLe Study team. Haemorrhoidal artery ligation versus rubber band ligation for the management of symptomatic second-degree and third-degree haemorrhoids (HubBLe): a multicentre, open-label, randomised controlled trial. Lancet. 2016 Jul 23;388(10042):356-364. doi: 10.1016/S0140-6736(16)30584-0. Epub 2016 May 25. PMID 27236344
- [Background] Fernandes V, Fonseca J. Polidocanol Foam Injected at High Doses with Intravenous Needle: The (Almost) Perfect Treatment of Symptomatic Internal Hemorrhoids. GE Port J Gastroenterol. 2019 May;26(3):169-175. doi: 10.1159/000492202. Epub 2018 Aug 31. PMID 31192285
- [Background] Lobascio P, Laforgia R, Novelli E, Perrone F, Di Salvo M, Pezzolla A, Trompetto M, Gallo G. Short-Term Results of Sclerotherapy with 3% Polidocanol Foam for Symptomatic Second- and Third-Degree Hemorrhoidal Disease. J Invest Surg. 2021 Oct;34(10):1059-1065. doi: 10.1080/08941939.2020.1745964. Epub 2020 Apr 15. PMID 32290709
- [Background] Forlini A, Manzelli A, Quaresima S, Forlini M. Long-term result after rubber band ligation for haemorrhoids. Int J Colorectal Dis. 2009 Sep;24(9):1007-10. doi: 10.1007/s00384-009-0698-y. Epub 2009 Apr 23. PMID 19387663
- [Background] Azizi R, Rabani-Karizi B, Taghipour MA. Comparison between Ultroid and rubber band ligation in treatment of internal hemorrhoids. Acta Med Iran. 2010 Nov-Dec;48(6):389-93. PMID 21287479
- [Background] Watson NF, Liptrott S, Maxwell-Armstrong CA. A prospective audit of early pain and patient satisfaction following out-patient band ligation of haemorrhoids. Ann R Coll Surg Engl. 2006 May;88(3):275-9. doi: 10.1308/003588406X98649. PMID 16719998
- [Background] Pol RA, van der Zwet WC, Hoornenborg D, Makkinga B, Kaijser M, Eeftinck Schattenkerk M, Eddes EH. Results of 244 consecutive patients with hemorrhoids treated with Doppler-guided hemorrhoidal artery ligation. Dig Surg. 2010;27(4):279-84. doi: 10.1159/000280020. Epub 2010 Jul 31. PMID 20689288
- [Background] Walega P, Romaniszyn M, Kenig J, Herman R, Nowak W. Doppler-guided hemorrhoid artery ligation with Recto-Anal-Repair modification: functional evaluation and safety assessment of a new minimally invasive method of treatment of advanced hemorrhoidal disease. ScientificWorldJournal. 2012;2012:324040. doi: 10.1100/2012/324040. Epub 2012 Apr 1. PMID 22547979
- [Background] Wilkerson PM, Strbac M, Reece-Smith H, Middleton SB. Doppler-guided haemorrhoidal artery ligation: long-term outcome and patient satisfaction. Colorectal Dis. 2009 May;11(4):394-400. doi: 10.1111/j.1463-1318.2008.01602.x. Epub 2008 Jun 28. PMID 18573116
- [Background] Alshreef A, Wailoo AJ, Brown SR, Tiernan JP, Watson AJM, Biggs K, Bradburn M, Hind D. Cost-Effectiveness of Haemorrhoidal Artery Ligation versus Rubber Band Ligation for the Treatment of Grade II-III Haemorrhoids: Analysis Using Evidence from the HubBLe Trial. Pharmacoecon Open. 2017 Sep;1(3):175-184. doi: 10.1007/s41669-017-0023-6. PMID 29441497
- [Derived] Neves S, Falcao D, Povo A, Castro-Pocas F, Oliveira J, Salgueiro P. 3% polidocanol foam sclerotherapy versus hemorrhoidal artery ligation with recto anal repair in hemorrhoidal disease grades II-III: a randomized, pilot trial. Rev Esp Enferm Dig. 2023 Mar;115(3):115-120. doi: 10.17235/reed.2022.8568/2022. PMID 35638762